CLINICAL TRIAL: NCT01213641
Title: An Open-label, Long-term, Prospective, Observational Study to Monitor the Safety and Effectiveness of Ilaris in CAPS Patients
Brief Title: Clinical Outcomes and Safety: A Registry Study of Ilaris (Canakinumab) Patients
Acronym: B-Confident
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CACZ885D2401
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Cryopyrin-associated Periodic Syndromes (CAPS); Familial Cold Autoinflam Syn (FCAS); Muckle-wells Syn (MWS); Neonatal Onset Multisystem Inflam Disease (NOMID)
Keywords: Cryopyrin-associated periodic syndromes(CAPS); CIAS1 protein; NLRP3 protein; human cryopyrin protein; Familial Cold Autoinflammatory Syndrome(FCAS); Muckle-Wells Syndrome(MWS); Neonatal Onset Multisystem Inflammatory disease(NOMID); NALP3; canakinumab; Interleukin-1(IL-1)
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this observational study is to collect additional information regarding long-term safety and effectiveness of Ilaris in the treatment of CAPS patients in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Ilaris (canakinumab) at the time of enrollment as part of medical care

Exclusion Criteria:

* Local regulations in some locations may exclude patients who receive Ilaris for a non-approved indication
* Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with CAPS and treated with canakinumab. Patients treated with canakinumab for other autoinflammatory diseases may be included where allowed per local regulations.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2009-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To monitor and further explore the overall safey of canakinumab focusing in serious infections | At least 5 years

SECONDARY OUTCOMES:
Long-term impact of Ilaris on disease progression (including systemic AA amyloidosis as evidenced by renal function, neurologic and ophthalmologic symptoms, and sensorineural deafness) | At least 5 years
Growth and development patterns of children aged 4 to 18 years of age exposed to Ilaris | at least 5 years
Identify previously unrecognized serious adverse drug reactions in the treated population | at least 5 years
Usage and patterns of dosing of Ilaris in routine clinical practice | at least 5 years
Incidence of serious infections | at least 5 years
Incidence of malignancies | at least 5 years
Incidence of hypersensitivity reactions | at least 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- United States (3):
  - Little Rock Allergy and Asthma Clinic, Little Rock, Arizona
  - Allergy Center at Brookstone, Columbus, Georgia
  - Rush Presbyterian - St. Lukes Medical Center, Chicago, Illinois
- Austria (2):
  - Novartis Investigative site, Bregenz
  - Novartis Investigative site, Vienna
- Germany (7):
  - Novartis Investigative site, Dresden
  - Novartis Investigative site, Hamburg
  - Novartis Investigative site, Heidelberg
  - Novartis Investigative site, Herne
  - Novartis Investigative site, Kiel
  - Novartis Investigative site, Schweinfurt
  - Novartis Investigative site, Tübingen
- Novartis Investigative site, Oslo, Norway
- Switzerland (4):
  - Novartis Investigative site, Aarau
  - Novartis Investigative site, Basel
  - Novartis Investigative site, Geneva
  - Novartis Investigative site, Lausanne

REFERENCES:
- [Derived] Walker UA, Tilson HH, Hawkins PN, Poll TV, Noviello S, Levy J, Vritzali E, Hoffman HM, Kuemmerle-Deschner JB; CACZ885D2401 Study Investigators. Long-term safety and effectiveness of canakinumab therapy in patients with cryopyrin-associated periodic syndrome: results from the beta-Confident Registry. RMD Open. 2021 May;7(2):e001663. doi: 10.1136/rmdopen-2021-001663. PMID 34001647